CLINICAL TRIAL: NCT01231464
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multi-Center Study to Evaluate the Efficacy and Safety of Fluticasone Furoate Nasal Spray for 2 Weeks in Chinese Adult and Adolescent Subjects With Allergic Rhinitis
Brief Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Fluticasone Furoate Nasal Spray for 2 Weeks in Chinese Adult and Adolescent Subjects With Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 113342
Record Dates: First submitted 2010-10-28; First posted 2010-11-01 (Estimated); Results first posted 2011-02-04 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-06

CONDITIONS: Rhinitis, Allergic, Perennial; Allergic Rhinitis
Keywords: safety; efficacy; placebo; allergic rhinitis; fluticasone furoate
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- placebo (Placebo Comparator): vehicle placebo nasal spray
  Interventions: Drug: placebo
- FFNS (Experimental): fluticasone furoate nasal spray
  Interventions: Drug: fluticasone furoate nasal spray

INTERVENTIONS:
Drug: fluticasone furoate nasal spray — fluticasone furoate nasal spray 110ug, once daily
  Arms: FFNS
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
The objective of this study is to compare the efficacy and safety of Fluticasone Furoate Nasal Spray (FFNS), that is FFNS with placebo in Chinese adult and adolescent subjects with Allergic Rhinitis as AR. There are 3 phases, 2 to14 day run in, 2 week treatment, and 3 to 5 day follow up. After run in period, at least 360 subjects with AR ( ages of 12yrs and 65yrs, inclusive) will be randomised to receive FFNS 110ug once daily or placebo for 2 weeks. The primary endpoint is the change from baseline of reflective total nasal symptom score (rTNSS) during treatment period, and the secondary endpoints include mean change from baseline in nasal finding scores by rhinoscopy at completion of study treatment, and severity of overall inference in activities of daily living. Safety measures include AE (Adverse Event) reports, ECGs (Electrocardiograph), physical exams, vital signs, and nasal exam. In addition, reflective total ocular symptom score (rTOSS) will be measured as an explorative endpoint, only in the specific AR (Allergic Rhinitis) patients with severe ocular symptoms.

DETAILED DESCRIPTION:
This is a multicenter, 2 week, double blind, randomized, placebo controlled trial. 7 investigational sites will be enlisted to randomize at least 360 subjects (outpatients) during 2009 and 2010. Throughout the entire study period, no antiallergy drugs and rhinitis medication, including rescue medication for symptom relief and anti-hyperactivity will be allowed. The run in period will consist of a minimum of 2 days and a maximum of 14 days. During this period, intermittent allergic rhinitis(IAR) or persistent allergic rhinitis(PER) should be diagnosed confirmatively as the definition from the current ARIA (Allergic Rhinitis and its Impact on Asthma) guideline and the coming effective Chinese allergic rhinitis management guideline. Subjects will assess their nasal symptom scores and compliance in dairy cards to confirm whether to meet randomization criteria. During the treatment period, subjects are randomized (1 and 1 ratio) to FFNS 110ug or matching vehicle placebo nasal spray to self administer intranasal treatment once daily for 2 weeks. Subjects will rate their nasal symptom scores and also document their study drug administration and compliance, any medication conditions experienced, and any concomitant medications taken in their dairy cards. Subjects also assess the severity of overall interference in activities of diary living(ADL) at baseline and the end of study treatment in their questionnaire. At baseline and the end of study treatment, investigators rate nasal findings scores by rhinoscopy, and record them in patient notes. A follow up telephone contact will be made 3 to 5 days after completion of study treatment/early withdrawal to assess for any post treatment adverse effects. The primary endpoint is the change from baseline of reflective total nasal symptom score(rTNSS) during treatment period, and the secondary endpoints include at completion of study treatment, mean change from baseline in nasal finding scores by rhinoscopy, and the severity of overall inference in activities of daily living. The safety measures include ECGs, vital exams, physical exams, and AE reports. In addition, reflective total ocular symptom score(rTOSS) will be measured as an explorative endpoint, only in the specific AR patients with severe ocular symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Subjects can be enrolled when meeting all criteria as below.

  1. Chinese adolescent and adult (male or eligible female) outpatients with the age of >=12 years
  2. Confirmative diagnosis of IAR or PER (as definitions from ARIA 2008 and the coming effective Chinese AR management guideline ), by medical history, symptoms, skin prick tests (SPTs)
  3. Subject must be symptomatic at screening and willing to maintain same environment throughout the study
  4. Ability to comply with study procedures
  5. Literate

Exclusion Criteria:

* Subjects should be excluded when meeting one of criteria as below.

  1. Having complications of nasal disease, or vasomotor rhinitis, rhinitis with eosinophilia, or drug rhinitis
  2. Having complications of bacterial/viral infection of upper respiratory tract
  3. Having significant systemic diseases
  4. History of hypersensitivity to steroids and ingredients
  5. Pregnant women or under lactation
  6. Patients who started, discontinued or changed dose of desensitization therapy within 30 days before visit 1
  7. Patients planning to travel outside the region
  8. Patients judged to be inappropriate by investigators
  9. Patients who participated in another study within 4 months before screening
  10. Patients who could not withdraw drugs during screening period or secure withdrawal period until the initiation day of administration, e.g.

      1. allergy medications
      2. other medications that may affect allergic rhinitis or its symptoms
      3. any medications that significantly inhibit CYP3A4, including ritonavir and ketoconazole

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2009-09; Primary Completion 2010-05 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- China (6):
  - GSK Investigational Site, Nanjing, Jiangsu
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Wuhan

REFERENCES:
- [Derived] Han D, Liu S, Zhang Y, Wang J, Wang D, Kong W, Wang S, Cheng L, Zhang L; Chinese Allergic Rhinitis Collaborative Research Group. Efficacy and safety of fluticasone furoate nasal spray in Chinese adult and adolescent subjects with intermittent or persistent allergic rhinitis. Allergy Asthma Proc. 2011 Nov-Dec;32(6):472-81. doi: 10.2500/aap.2011.32.3474. Epub 2011 Aug 31. PMID 21888757

RESULTS

PARTICIPANT FLOW:
Groups:
- FFNS 110 mcg: Fluticasone Furoate Nasal Spray (FFNS) 110 micrograms (mcg) once daily (QD)
- Placebo: Matching Vehicle Placebo Nasal Spray QD
Period: Overall Study
Arm/Group | FFNS 110 mcg | Placebo
Started | 182 | 183
Completed | 177 | 176
Not Completed | 5 | 7
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 1 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FFNS 110 mcg | Placebo | Total
Number analyzed (Participants) | 181 | 182 | 363
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline characteristics are summarized for the Full Analysis Set (FAS), comprised of all participants who were randomized and received at least one dose of study medication.
  Years | 31.8 (10.72) | 33.0 (10.95) | 32.4 (10.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 99 | 196
  Male | 84 | 83 | 167
Race/Ethnicity, Customized [Number; unit: participants]
  Chinese | 181 | 182 | 363
  Not Chinese | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline Over the Entire Treatment Period in the Daily Reflective Total Nasal Symptom Score (rTNSS)
Description: The Total Nasal Symptom Score (TNSS; possible score of 0-12) is the sum of 4 individual participant-assessed symptom scores for rhinorrhea, nasal congestion, nasal itching, and sneezing, each evaluated using a scale of 0=None, 1=Mild, 2=Moderate, or 3=Severe. The rTNSS was performed in the morning (AM rTNSS) and evening (PM rTNSS) and assessed the participant's symptoms over the preceding 12 hours. The daily rTNSS is the average of the AM rTNSS and PM rTNSS assessments. Mean changes from baseline over the entire treatment period were calculated as treatment period rTNSS minus baseline rTNSS.
Time Frame: Baseline through entire treatment period (Day 1 through Day 14)
Population: Full Analysis Set (FAS): all participants who were randomized and received at least one dose of study medication. Only participants for whom both baseline and post-baseline data were available were included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: Points on a scale
Arm/Group | FFNS 110 mcg | Placebo
Number analyzed (Participants) | 179 | 178
Points on a scale | -4.226 (0.1646) | -2.728 (0.1656)
Statistical Analysis 1: Comparison: FFNS 110 mcg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean Difference = -1.498, 95% CI 2-sided [-1.897 to -1.009] — Besides treatment, the ANCOVA analysis also adjusted for baseline, center, gender, age, and classification of AR (Intermittent Allergic Rhinitis [IAR] or Persistent Allergic Rhinitis [PER])

2. Secondary Outcome: Mean Change From Baseline (Visit 2) to the End of Study (Visit 4/Early Withdrawal) in Nasal Finding Score by Rhinoscopy
Description: The nasal finding score by rhinoscopy (possible score of 0-12) is the sum of 4 individual investigator assessed scores for swelling of inferior nasal concha mucosa, color of inferior nasal concha mucosa, watery secretion volume, and description of rhinorrhea. The symptoms were assessed using a scale of 0=None, 1=Mild, 2=Moderate, 3=Severe. Mean change from baseline to the end of study in nasal finding score by rhinoscopy was calculated as the nasal finding score by rhinoscopy at Visit 4/Early Withdrawal minus the nasal final finding score by rhinoscopy at Visit 2.
Time Frame: Baseline through end of study (Day 1 through Day 15/Early Withdrawal)
Population: FAS Population. Only participants for whom both baseline and post-baseline data were available were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Points on a scale
Arm/Group | FFNS 110 mcg | Placebo
Number analyzed (Participants) | 176 | 177
Points on a scale | -4.2 (0.22) | -2.9 (0.22)

3. Secondary Outcome: Mean Change From Baseline (Visit 2) to the End of Study (Visit 4/Early Withdrawal) in Severity of Overall Interference in Activities of Daily Living
Description: The severity of overall interference in activities of daily living at baseline and the end of study was assessed by the investigator on the scale of 0=None, 1=Mild, 2=Moderate, 3=Severe. The mean change from baseline to the end of study in severity of overall interference in activities of daily living was calculated as the severity of overall interference in activities of daily living at Visit 4/Early Withdrawal minus severity of overall interference in activities of daily living at Visit 2.
Time Frame: Baseline through end of study (Day 1 through Day 15/Early Withdrawal)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Points on a scale
Groups:
- FFNS 110 mcg: Fluticasone Furoate Nasal Spray (FFNS) 110 micrograms (mg) once daily (QD)
Arm/Group | FFNS 110 mcg | Placebo
Number analyzed (Participants) | 160 | 165
Points on a scale | -1.2 (0.07) | -0.8 (0.07)

ADVERSE EVENTS:
Description: Serious and non-serious adverse events were collected in the Safety Set, comprised of all participants who were randomized and received at least one dose of study medication.
Arm/Group | FFNS 110 mcg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/181 | 0/182
Other Adverse Events (participants affected / at risk) | 13/181 | 9/182
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FFNS 110 mcg (N=181) | Placebo (N=182)
Upper respiratory tract infection (Infections and infestations) | 4 | 2
Nasopharyngitis (Infections and infestations) | 0 | 3
Oral herpes (Infections and infestations) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sputum (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 0 | 1
Blood urine present (Investigations) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.